CLINICAL TRIAL: NCT04576923
Title: Quantitative Ultrasound With Liver Incytes for Evaluation of Non-Alcoholic Fatty Liver Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of coordinator resources
Sponsor: Indiana University (Other)
Collaborators: Sonic Incytes (Industry)
Responsible Party: Principal Investigator, Samer Gawrieh, Professor of Clinical Medicine, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Liver Incytes for NAFLD; 2009698457 (Other: Indiana University IRB)
Record Dates: First submitted 2020-09-30; First posted 2020-10-06 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: NAFLD; NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: All participants will undergo quantitative ultrasound with Liver Incytes by a certified technician.
Masking Description: This is an open label study in that all participants will receive the same study procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Velacur by Sonic Incytes (Experimental): Patients with known or suspected Non-Alcoholic Fatty Liver Disease (NAFLD) or Non-Alcoholic Steatohepatitis (NASH) will be scanned with Velacur for assessment of liver fibrosis.
  Interventions: Diagnostic Test: Velacur by Sonic Incytes

INTERVENTIONS:
Diagnostic Test: Velacur by Sonic Incytes — liver stiffness measurement

SUMMARY:
The purpose of this study is to prospectively evaluate the utility of Liver Incytes in assessing NAFLD with or without advanced fibrosis in patients seen in liver clinics for suspected NAFLD diagnosis.

DETAILED DESCRIPTION:
The proposed study will evaluate the performance characteristics of LSM as a measure of fibrosis and ACE as a measure of hepatic steatosis by Liver Incytes in patients with different stages of NAFLD. In addition, the diagnostic accuracy of ACE will be compared to CAP and LSM as measured by Liver Incytes to that measured by FibroScan® using liver histology as the reference standard. The performance of these two methods will also be compared to that of non-invasive blood based markers such as APRI, FIB4, and NAFLD fibrosis score in predicting advanced fibrosis in biopsy proven NAFLD.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 21 years or older
2. Suspected NAFLD or NASH with plans to undergo standard of care liver biopsy
3. History of biopsy proven NAFLD or NASH within 6 months prior to enrollment
4. Planned liver biopsy for evaluation of NAFLD within 6 months of enrollment
5. Ability to provide informed consent

Exclusion Criteria:

1. Fasting for less than three hours prior to the scan
2. Subject is a pregnant or lactating female
3. Subject with current, significant alcohol consumption or history of significant alcohol consumption for a period of more than 3 consecutive months any time within 1 year prior to screening. Significant alcohol consumption is defined as more than 20 gram per day in females and more than 30 grams per day in males, on average (a standard drink in the US is considered to be 14 grams of alcohol).
4. Subject is unable to reliably quantify alcohol consumption based upon local study physician judgment.
5. Subject uses drugs historically associated with NAFLD (amiodarone, methotrexate, systemic glucocorticoids, tetracyclines, tamoxifen, estrogens at doses greater than those used for hormone replacement, anabolic steroids, valproic acid, and other known hepatotoxins) for more than 2 weeks in the year prior to screening
6. Subject with history of cirrhosis or clinical evidence of hepatic decompensation as defined by the presence of any of the following abnormalities at screening

   1. Serum albumin less than 3.5 grams/deciliter (g/dL).
   2. INR greater than 1.5.
   3. Direct bilirubin greater than 1.3 milligrams per deciliter (mg/dL).
7. Subject has a history of bleeding esophageal varices, ascites or hepatic encephalopathy
8. Subject has history of other forms of chronic liver diseases such as viral hepatitis, autoimmune hepatitis, cholestatic liver disease (primary biliary cirrhosis or primary sclerosing cholangitis).
9. Subject with active substance abuse
10. Acute hepatitis defined as AST/ALT > 500 U/L
11. Patients with a pacemaker or defibrillator
12. Ascites

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samer Gawrieh, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Division of Gastroenterolgy and Hepatology, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 36 participants who enrolled in the study, only 21 people had a valid Velacur study and valid ultrasound elasticity imaging. All 36 people completed the study but 15 people were later found to have results that were deemed to not be valid upon review by Sonic Incytes.
Pre-assignment Details: Of the 36 participants who enrolled in the study, only 21 people had a valid Velacur study and valid ultrasound elasticity imaging. All 36 people completed the study but 15 people were later found to have results that were deemed to not be valid upon review by Sonic Incytes.
Groups:
- Velacur by Sonic Incytes: Patients with known or suspected Non-Alcoholic Fatty Liver Disease (NAFLD) or Non-Alcoholic Steatohepatitis (NASH) will be scanned with Liver Incytes.
  Of the 36 participants who enrolled in the study, only 21 people had a valid Velacur study and valid ultrasound elasticity imaging. All 36 people completed the study but 15 people were later found to have results that were deemed to not be valid upon review by Sonic Incytes.
Period: Overall Study
Arm/Group | Velacur by Sonic Incytes
Started | 36
Completed | 21
Not Completed | 15
Not completed — 15 had scans that were determined to be invalid and these are not reported within the results. | 15

BASELINE CHARACTERISTICS:
Population: A total of 21 people underwent both Velacur and transient elastography via FibroScan and had results considered to be reliable.
Arm/Group | Velacur by Sonic Incytes
Number analyzed (Participants) | 21
Age, Continuous [Median (Standard Deviation); unit: years] | 58 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 21
BMI measured in kg/m^2 [Mean (Standard Deviation); unit: kg/m^2] | 34.4 (7.4)

OUTCOME MEASURES:

1. Primary Outcome: Liver Stiffness Measured by Velacur
Description: Assessing correlation of liver stiffness measurements (LSM) as measured by Velacur to grade of fibrosis on liver histology of patients with NAFLD who underwent standard of care liver biopsy. Results are reported per fibrosis category: F0, F1, F2, F3, and F4.
Time Frame: one day
Population: Of the 36 enrolled participants, 21 were determined to have results that were considered to be reliable for both the Velacur and transient elastography via FibroScan and underwent a liver biopsy less than 6 months prior to the Velacur and FibroScan measurements.
  Results are reported for two participants with F0 biopsy results.
Measure: Median (Standard Deviation); unit: kPa
Groups:
- Velacur by Sonic Incytes for Stage F0: Patients with known or suspected Non-Alcoholic Fatty Liver Disease (NAFLD) or Non-Alcoholic Steatohepatitis (NASH) will be scanned with Velacur and FibroScan and results will be compared to historical liver biopsy results. Liver biopsy was completed within 6 months of the Velacur and Fibroscan measurements.
  Results are reported for each group as determined by staging on liver biopsy: F0
- Velacur by Sonic Incytes for Stage F1: Patients with known or suspected Non-Alcoholic Fatty Liver Disease (NAFLD) or Non-Alcoholic Steatohepatitis (NASH) will be scanned with Velacur and FibroScan and results will be compared to historical liver biopsy results. Liver biopsy was completed within 6 months of the Velacur and Fibroscan measurements.
  Results are reported for each group as determined by staging on liver biopsy: F1
- Velacur by Sonic Incytes for Stage F2: Patients with known or suspected Non-Alcoholic Fatty Liver Disease (NAFLD) or Non-Alcoholic Steatohepatitis (NASH) will be scanned with Velacur and FibroScan and results will be compared to historical liver biopsy results. Liver biopsy was completed within 6 months of the Velacur and Fibroscan measurements.
  Results are reported for each group as determined by staging on liver biopsy: F2
- Velacur by Sonic Incytes for Stage F3: Patients with known or suspected Non-Alcoholic Fatty Liver Disease (NAFLD) or Non-Alcoholic Steatohepatitis (NASH) will be scanned with Velacur and FibroScan and results will be compared to historical liver biopsy results. Liver biopsy was completed within 6 months of the Velacur and Fibroscan measurements.
  Results are reported for each group as determined by staging on liver biopsy: F3
- Velacur by Sonic Incytes for Stage F4: Patients with known or suspected Non-Alcoholic Fatty Liver Disease (NAFLD) or Non-Alcoholic Steatohepatitis (NASH) will be scanned with Velacur and FibroScan and results will be compared to historical liver biopsy results. Liver biopsy was completed within 6 months of the Velacur and Fibroscan measurements.
  Results are reported for each group as determined by staging on liver biopsy: F4
Arm/Group | Velacur by Sonic Incytes for Stage F0 | Velacur by Sonic Incytes for Stage F1 | Velacur by Sonic Incytes for Stage F2 | Velacur by Sonic Incytes for Stage F3 | Velacur by Sonic Incytes for Stage F4
Number analyzed (Participants) | 2 | 4 | 5 | 5 | 5
kPa | 9.8 (4.4) | 7.2 (2.3) | 7.4 (1.6) | 7.5 (1.9) | 10.5 (5.0)

2. Primary Outcome: Liver Stiffness Measured by Transient Elastography
Description: Assessing correlation of liver stiffness measurements (LSM) as measured by FibroScan to grade of fibrosis on liver histology of patients with NAFLD who underwent standard of care liver biopsy. Results are reported per fibrosis category: F0, F1, F2, F3, and F4.
Time Frame: one day
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: kPa
Arm/Group | Velacur by Sonic Incytes for Stage F0 | Velacur by Sonic Incytes for Stage F1 | Velacur by Sonic Incytes for Stage F2 | Velacur by Sonic Incytes for Stage F3 | Velacur by Sonic Incytes for Stage F4
Number analyzed (Participants) | 2 | 4 | 5 | 5 | 5
kPa | 11.1 (4.3) | 10.1 (3.5) | 15.3 (8.3) | 7.5 (1.9) | 18.2 (9.1)

3. Other Pre Specified Outcome: Correlation of Velacur Measurements to Non-Invasive Blood Markers for Predicting Advanced Fibrosis
Description: This was initially included in our study protocol as an outcome measurement. However, we realized that these markers were not being routinely collected and the data are simply not available. Therefore, no outcome data are or can be included for this measurement.
Time Frame: one day
Population: During the conduct of this trial, we realized that these markers were not being routinely collected. For this study, no data for these markers were collected and are thus not available. As a result, no outcome data are or can be included for this measurement for any of the stages.
Arm/Group | Velacur by Sonic Incytes for Stage F0 | Velacur by Sonic Incytes for Stage F1 | Velacur by Sonic Incytes for Stage F2 | Velacur by Sonic Incytes for Stage F3 | Velacur by Sonic Incytes for Stage F4
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of study participation. This is a minimal risk study with only one study visit lasting less than one hour.
Description: The definition of adverse event utilized in this trial correlates with the clincialtrials.gov definition of adverse events.
Groups:
- Velacur by Sonic Incytes: Patients with known or suspected Non-Alcoholic Fatty Liver Disease (NAFLD) or Non-Alcoholic Steatohepatitis (NASH) will be scanned with Liver Incytes.
  Of the 36 participants who enrolled in the study, only 21 people had a valid Velacur study and valid ultrasound elasticity imaging. All 36 people completed the study but 15 people were later found to have results that were deemed to not be valid upon review by Sonic Incytes.
  Adverse events were collected for the duration of study participation. This is a minimal risk study with only one study visit lasting less than one hour.
Arm/Group | Velacur by Sonic Incytes
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/23/NCT04576923/Prot_006.pdf
  • Statistical Analysis Plan (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/23/NCT04576923/SAP_007.pdf